CLINICAL TRIAL: NCT04007250
Title: FENIX™ Continence Restoration System Registry
Status: Completed | Type: Observational
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 3422
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Fecal Incontinence; Faecal Incontinence
Keywords: Magnetic Anal Sphincter Augmentation; FENIX™ continence restoration system; Magnetic Anal Sphincter
MeSH Terms: conditions — Fecal Incontinence; Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- FENIX participants: Individuals being treated with the FENIX™ Continence Restoration System.
  Interventions: Device: FENIX™ Continence Restoration System

INTERVENTIONS:
Device: FENIX™ Continence Restoration System — The FENIX™ Continence Restoration System is indicated for use for the treatment of chronic fecal incontinence in patients who have failed or are not candidates for more conservative therapy. The FENIX™ System Implant is placed around the external anal sphincter to augment a weak anal sphincter and restore continence.
  The FENIX™ System is comprised of the following components:
  * FENIX™ System Implant
  * FENIX™ System Anal Sphincter Sizing Tool The FENIX™ System Implant consists of a series of titanium beads with magnetic cores that are connected with independent titanium wires to form an annular shape. The attractive force of the magnetic beads is designed to provide additional strength to keep a weak anal sphincter closed.
  Other Names: Magnetic anal sphincter augmentation

SUMMARY:
The FENIX Registry is a multi-center, observational database designed to collect data regarding the FENIX™ Continence Restoration System in everyday clinical practice, evaluate the clinical course of patients from pre-operative assessment through five years post-surgery and Track and monitor effectiveness and safety through the use of a bowel diary, fecal incontinence quality-of-life measures and adverse event reporting. Up to 25 sites will participate in the Registry. Sites to enroll consecutive eligible patients into the Registry. Registry will enroll approximately 200 FENIX patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals being treated with the FENIX™ Continence Restoration System
* Individuals who have provided appropriate authorization per institutional policy and procedure to have clinical and health information collected for the FENIX Registry.
* Individuals willing to complete a 14-day bowel diary, questionnaires and comply with all required follow-up.

Exclusion Criteria:

* Known circumstances that would make it unlikely for an individual to complete the five-year follow-up (e.g. life expectancy <5 years)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Chronic fecal incontinence patients who have failed or are not candidates for more conservative therapy.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2012-01-07 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Change in fecal incontinence (FI) episodes | Evaluate at 6 months and then annually at 12 months through 60 months post implant
  Proportion of participants with at least a 50% reduction in FI episodes per week
Change in fecal incontinence days | Evaluate at 6 months and then annually at 12 months through 60 months post implant
  Proportion of participants achieving at least 50% reduction in FI days per week and urgent episodes
Adverse events related to the FENIX system | assessed up to last follow up [max 60 months]
  From the time of implant and at each follow-up visit, safety will be evaluated by characterizing adverse events (AEs) related to the FENIX system and summarizing incidence rates. Serious device-related AEs will be summarized separately.
Change in Fecal Incontinence Quality of Life: Fecal Incontinence Quality of Life (FIQOL) score. | Evaluate at 6 months and then annually at 12 months through 60 months post implant
  Proportion of patients with improvement in Fecal Incontinence Quality of Life (FIQOL) score. The Fecal Incontinence Quality of Life Scale consists of 29 items divided into 4 scales:
  * Lifestyle (10 items)
  * Coping/Behavior (9 items)
  * Depression/Self Perception (7 items)
  * Embarrassment (3 items) Scales range from 1 to 5, scale scores are the average (mean) of all responses to all items in each scale. A lower score indicated a lower quality of life. The scales are not combined for a "composite" or total score but always presented individually.

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital of Nantes, Nantes, France
- Kliniken Essen-Mitte, Essen, Germany

IPD SHARING:
Plan to Share IPD: No